CLINICAL TRIAL: NCT06039982
Title: Establish a New Noninvasive Diagnostic Model Based on Clinical Indicators to Evaluate the Vaginal Invasion in Cervical Cancer Patients
Brief Title: A Diagnostic Nomogram for Predicting Vaginal Invasion in Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Yang Sun
Record Dates: First submitted 2023-09-11; First posted 2023-09-15 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cervix Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cervical cancer treated with surgery: The inclusion criteria were: (1) pathologically confirmed CC; (2) FIGO stage IB-IIA according to the result of physical examination and imaging; (3) abdominal MRI was performed within three weeks before surgery. Exclusion criteria were: (1) accompanied with other tumors. (2) with chronic infectious disease. (3) incomplete clinical data.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to develop a diagnostic nomogram based on clinical factors with the prediction values of vaginal invasion in cervical cancer to optimize the treatment plan and surgical procedures.

DETAILED DESCRIPTION:
Vaginal invasion is a crucial index participant in cervical cancer tumor staging and prognosis prediction. However, the roles of vaginal invasion are overlooked in the literature, compared with those of lymph node metastasis and parametrial invasion. As far as we know, this study is novel to construct a nomogram to predict the probability of pathologic vaginal invasion occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cervical cancer;
* FIGO2018 stage IB-IIA according to the result of physical examination and images;
* No preoperative treatment before surgery;
* Abdominal MRI is performed within three weeks before surgery. Blood routine, biochemistry, blood tumor markers and coagulation function were examined within 1 week before surgery.
* All patients undergo radical hysterectomy (RH) with bilateral pelvic lymphadenectomy or paraaortic lymph node dissection.

Exclusion Criteria:

* Accompanied with other tumors;
* Accompanied with chronic infectious and immune diseases;
* Incomplete clinical data.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we collect the medical data of cervical cancer patients in Fujian Cancer Hospital. All patients received a standardized staging evaluation before radical hysterectomy with bilateral pelvic lymphadenectomy, preoperative laboratory tests, abdominal MRI/CT, and thoracic CT.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
vaginal invasion | 7 days after surgery
  100 cervical cancer patients who underwent radical hysterectomy (RH) with bilateral pelvic lymphadenectomy were pathologically assessed for vaginal invasion. The primary outcome is vaginal invasion or no-vaginal invasion. Pathological vaginal invasion is defined as cervix tumor disruption of the vaginal wall.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvo G, Odetto D, Saez Perrotta MC, Noll F, Perrotta M, Pareja R, Wernicke A, Ramirez PT. Measurement of tumor size in early cervical cancer: an ever-evolving paradigm. Int J Gynecol Cancer. 2020 Aug;30(8):1215-1223. doi: 10.1136/ijgc-2020-001436. Epub 2020 Jul 6. PMID 32636272
- [Background] Thomeer MG, Gerestein C, Spronk S, van Doorn HC, van der Ham E, Hunink MG. Clinical examination versus magnetic resonance imaging in the pretreatment staging of cervical carcinoma: systematic review and meta-analysis. Eur Radiol. 2013 Jul;23(7):2005-18. doi: 10.1007/s00330-013-2783-4. Epub 2013 Mar 1. PMID 23455762
- [Background] Wagner-Larsen KS, Lura N, Salvesen O, Halle MK, Forsse D, Trovik J, Smit N, Krakstad C, Haldorsen IS. Interobserver agreement and prognostic impact for MRI-based 2018 FIGO staging parameters in uterine cervical cancer. Eur Radiol. 2022 Sep;32(9):6444-6455. doi: 10.1007/s00330-022-08666-x. Epub 2022 Mar 24. PMID 35332408